CLINICAL TRIAL: NCT03312179
Title: STEMI and Mutlivessels Coronary Artery Stenosis: Effect of Incretin Treatment
Brief Title: STEMI and Incretins Treatment
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, MD, MSc, PHD, University of Campania Luigi Vanvitelli
Other Study IDs: 9/2017
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: STEMI; Coronary Artery Disease; Coronary Syndrome; Coronary Arteriosclerosis; Diabetes
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease; Angina, Unstable; Diabetes Mellitus | interventions — Percutaneous Coronary Intervention; Incretins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- diabetics STEMI: Diabetics patients admitted for ST elevation myocardial infarction (STEMI) and associated with multi vessels (Mv) non obstructive coronary artery stenosis (NOCS). These patients received percutaneous coronary intervention (PCI), and primary stenting (DES) of culprit lesion. Then these patients received full medical STEMI therapy.
  Interventions: Device: PCI and DES stenting
- non diabetics STEMI: Non diabetics patients admitted for ST elevation myocardial infarction (STEMI) and associated with multi vessels coronary artery stenosis(Mv) non obstructive coronary artery stenosis (NOCS). These patients received percutaneous coronary intervention (PCI), and primary stenting (DES) of culprit lesion. Then these patients received full medical STEMI therapy.
  Interventions: Device: PCI and DES stenting
- diabetics incretin-users STEMI: Diabetics patients admitted for ST elevation myocardial infarction (STEMI) and associated with multi vessels coronary artery stenosis (Mv) non obstructive coronary artery stenosis (NOCS). These patients received percutaneous coronary intervention (PCI), and primary stenting (DES) of culprit lesion. Then these patients received full medical STEMI therapy. These patients were treated by incretin therapy at last 6 months before study enrollment.
  Interventions: Device: PCI and DES stenting; Drug: Incretins
- diabetics never-incretin-users STEMI: Diabetics patients admitted for ST elevation myocardial infarction (STEMI) and associated with multi vessels coronary artery stenosis (Mv) non obstructive coronary artery stenosis (NOCS). These patients received percutaneous coronary intervention (PCI), and primary stenting (DES) of culprit lesion. Then these patients received full medical STEMI therapy. These diabetic patients were never treated by incretin therapy before study enrollment.
  Interventions: Device: PCI and DES stenting

INTERVENTIONS:
Device: PCI and DES stenting — Percutaneous coronary intervention (PCI) and direct stenting (DES) of culprit lesion vessel.
Drug: Incretins — Patients treated before study enrollment by incretin drugs (6 months drugs exposure)
  Groups: diabetics incretin-users STEMI

SUMMARY:
ST elevation myocardial infarction (STEMI) patients affected by multivessels coronary artery stenosis, represent a clinical relevant problem. The management and prognosis of these patents are supported by few literature data. Therefore, in this study authors enrolled real world diabetic vs. non diabetic patients admitted for STEMI and associated to multi vessels coronary disease. Then these diabetics were divided in incretin users (6 months of incretin treatment before study enrollment) vs. never incretin users. In these patients authors studied all cause mortality, cardiac mortality, and major adverse cardiac events at 12 months follow up.

DETAILED DESCRIPTION:
ST elevation myocardial infarction (STEMI) patients affected by multivessels coronary artery stenosis represent a class of patients really challenging to treat. In fact, treatment, clinical management, and prognosis are supported by few literature data. Therefore, in this study authors enrolled real world patients admitted for STEMI and associated to multi vessels coronary disease. Multivessels (Mv) coronary stenosis were characterized by non obstructive coronary stenosis (NOCS) as coronary lesions <50% with fractional flow reserve > 0.8. Therefore, STEMI was treated by percutaneous coronary intervention by primary angioplasty and direct stenting (DES stenting) of culprit vessel lesion. Then these STEMI-Mv-NOCS patients were divided in diabetics vs. non diabetics, and received conventional full medical therapy for STEMI. Then these diabetics were divided in incretin users (6 months of incretin treatment before study enrollment) vs. never incretin users. Study outcomes were all cause mortality, cardiac mortality, and major adverse cardiac events at 12 months follow up. Authors studied these study outcomes comparing diabetics vs. non diabetics at 12 moths follow up, and diabetics incretin-users vs. never-incretin-users.

ELIGIBILITY:
Inclusion Criteria:

aged >18, first STEMI, STEMI with multi vessels coronary stenosis.

Exclusion Criteria:

aged < 18, renal impairment, mono vessel STEMI, severe depression of left ventricle ejection fraction (LVEF <35%).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetics and non diabetics patients admitted for STEMI. In this population authors selected STEMI patients with multivessel (Mv) non obstructive coronary diseases (NOCS). These STEMI-Mv-NOCS had coronary lesions and stenosis <50%, with fractional flow reserve >0.8. In diabetics authors selected incretin users (6 months of incretin treatment before study enrollment) vs never-incretin-users diabetics.
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
all cause deaths | 12 months
  at 12 months follow up authors monitored and reported all cause mortality
cardiac deaths | 12 months
  at 12 months follow up authors monitored and reported mortality events due to cardiac causes
MACE | 12 months
  authors monitored and reported at follow up major adverse cardiac events (MACE): re-STEMI, NSTEMI, unstable angina, arrhythmias, stroke etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided